CLINICAL TRIAL: NCT04058613
Title: Effects of Maintaining Steady Albumin Levels by Targeted Albumin Therapy (TAT 4) on Survival and Liver Related Complications in Cirrhosis With Ascites and Low Serum Albumin Level- a Randomized Controlled Trial
Brief Title: Effects of Maintaining Steady Albumin Levels (TAT 4) on Survival and Liver Related Complications in Cirrhosis With Ascites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Shasthry SM, Associate Professor, Institute of Liver and Biliary Sciences, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ILBS-TAT4-01
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — ALB protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin (Experimental): Albumin infusions will be given at a dose of 40 g twice weekly till a steady albumin level of 4.0g/dl is reached followed by 100ml of 20% albumin at least once in two weeks to maintain a steady albumin level of 4.0g/dl along with the standard medical therapy
  Interventions: Drug: ALB Protein, Human
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ALB Protein, Human — Albumin infusions will be given at a dose of 40 g twice weekly till a steady albumin level of 4.0g/dl is reached followed by 100ml of 20% albumin at least once in two weeks to maintain a steady albumin level of 4.0g/dl along with the standard medical therapy
  Arms: Albumin
Other: placebo — placebo
  Arms: Placebo

SUMMARY:
Investigators intend to assess the utility of regular albumin infusions to maintain a targeted serum albumin level of 4.0 g/dl in newly detected cirrhotic patients with low albumin levels (<2.8g/dl) with ascites.

DETAILED DESCRIPTION:
Cirrhosis is characterized by progressive deterioration in liver functions. Liver's synthetic functions are inferred by serum albumin and INR estimation. Lower albumin level is a marker of severe liver disease and probability of worsening ascites, hepatorenal syndrome with increased risk for infections. Of the three recent RCTs on utility of long-term administration of albumin, two showed improvement in survival. The studies had included different patient populations (diuretic refractory ascites, high dose diuretics and patients on liver transplant waiting list) with different albumin infusion protocols and different end-points. These studies were done in advanced cases of cirrhosis. There is limited data on the utility of regular albumin infusions in early hepatic decompensation (albumin levels-<2.8g/dl with ascites) and the effect of maintaining a targeted albumin level on survival or liver related side effects. Investigators are trying to address this issue by starting regular albumin infusions at an earlier stage of liver decompensation.

ELIGIBILITY:
Inclusion Criteria:

* Newly detected cirrhotic patients aged more than 18 years
* Cirrhosis deﬁned by standard clinical, analytical and/or histological criteria
* Serum albumin level < 2.8g/dl with or without ascites
* Who would agree to give written informed consent

Exclusion Criteria:

* Uncontrolled HTN (sys>150/ dis >90 mmHg) or h/o any drug therapy for HTN
* Prior h/o Transjugular Intrahepatic Portosystemic Shunt (TIPS)
* Hepatocellular Carcinoma
* Active alcohol abuse within 3 months
* Patients presenting as Acute on Chronic Liver Failure
* Extrahepatic organ failure
* Known case of chronic heart failure or respiratory failure
* Diagnosed Chronic Kidney Disease
* Patients with hydrothorax
* Prior liver transplant recipient
* Human Immunodeficiency Virus infection
* Use of albumin infusion in the last one month
* CTP>12, MELD>28
* Total Bilirubin >3 g/dl
* Overt Hepatic Encephalopathy at Presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2019-09-10 (Estimated); Primary Completion 2020-08-08 (Estimated); Study Completion 2021-08-08 (Estimated)

PRIMARY OUTCOMES:
Transplant/Transintrahepatic Portosystemic Shunt (TIPS) free survival in both groups | 12 months
  1 year survival

SECONDARY OUTCOMES:
New onset refractory ascites in both the groups | 12 months
  refractory ascites is defined as non response to maximum tolerated dose of diuretics
Spontaneous bacterial peritonitis [SBP] in both groups | 12 months
  Spontaneous bacterial peritonitis is defined as ascitic fluid absolute neutrophil count > 250/ mL with or without culture positivity
Renal impairment in both groups | 12 months
  serum creatinine concentration >1•5 mg/dL
Hepatorenal Syndrome in both groups | 12 months
  Hepatorenal Syndrome type 1 is defined as new onset increase in serum creatinine level by 0.3 mg/dL or 50% increase from baseline
Hepatic encephalopathy grade 3 or 4 in both groups | 12 months
  HE as per West Haven criteria
Number of new cases with gastrointestinal bleeding in both groups | 12 months
  gastrointestinal bleeding as confirmed by endoscopic/clinical evidence of variceal bleed.
Requirement of paracentesis in both groups | 12 months
  Ascitic tapping for relieve of pressure symptoms or diagnosis of SBP
Requirement of diuretics in both groups | 12 months
  Frusemide or Aldactone for management of ascites
Number of hospitalizations per subject in both groups | 12 months
  Need for any cause hospitalization
New onset breathlessness/ Hypertension within 24 hours of albumin infusion in both groups | within 24 hours
  Development of cardiac overload
Quality of life by Ascite-Q questionnaire in both groups | 12 months
  semiquantitative questionnaire to be answered by the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India